CLINICAL TRIAL: NCT01669239
Title: OptiHER-Heart: A Prospective, Multicenter, Single-arm, Phase II Study to Evaluate the Safety of Neoadjuvant Liposomal Doxorubicin (Myocet®) Plus Paclitaxel, Trastuzumab, and Pertuzumab in Patients With HER2-positive Breast Cancer
Brief Title: Study of Neoadjuvant Myocet®, Paclitaxel, Pertuzumab, and Trastuzumab in HER2-positive Breast Cancer
Acronym: Opti-HER
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SOLTI Breast Cancer Research Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SOLTI-1002; 2012-001201-24 (EudraCT Number)
Record Dates: First submitted 2012-08-09; First posted 2012-08-20 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; HER2 positive; Neoadjuvant; Liposomal doxorubicin; Paclitaxel; Trastuzumab; Pertuzumab; Safety
MeSH Terms: conditions — Breast Neoplasms | interventions — liposomal doxorubicin; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Liposomal Doxorubicin (Experimental): Six cycles of:
  * Trastuzumab 4 mg/kg loading dose on Day 1 of the first cycle, then 2 mg/kg on Days 8 and 15 of the first cycle and on Days 1, 8, and 15 of the subsequent cycles, every 3 weeks
  * Pertuzumab 840 mg loading dose on Day 1 of the first cycle, then 420 mg on Day 1, every 3 weeks
  * Liposomal doxorubicin 50 mg/m2 on Day 1, every 3 weeks
  * Paclitaxel 80 mg/m2 on Days 1, 8, and 15, every 3 weeks
  Interventions: Drug: Liposomal Doxorubicin

INTERVENTIONS:
Drug: Liposomal Doxorubicin — Six cycles of:
  * Trastuzumab 4 mg/kg loading dose on Day 1 of the first cycle, then 2 mg/kg on Days 8 and 15 of the first cycle and on Days 1, 8, and 15 of the subsequent cycles, every 3 weeks
  * Pertuzumab 840 mg loading dose on Day 1 of the first cycle, then 420 mg on Day 1, every 3 weeks
  * Liposomal doxorubicin 50 mg/m2 on Day 1, every 3 weeks
  * Paclitaxel 80 mg/m2 on Days 1, 8, and 15, every 3 weeks
  Other Names: Myocet® (liposome-encapsulated doxorubicin)

SUMMARY:
This is a prospective, multicenter, single-arm, phase II study to evaluate the safety of neoadjuvant liposomal doxorubicin plus paclitaxel, trastuzumab, and pertuzumab in patients with HER2-positive breast cancer

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent for all study procedures according to local regulatory requirements prior to beginning specific protocol procedures
* Female patients
* Age 18-74 years
* ECOG Performance Status of 0 or 1
* Histologically confirmed, untreated, invasive breast carcinoma stage II-IIIB
* Tumor size > 2 cm by clinical or radiological assessment
* HER2+ invasive BC according to ASCO/CAP guidelines
* Known hormone receptor status or the possibility of its assessment
* Adequate organ function defined as:

  * Absolute Neutrophil Count (ANC) ≥ 1.5 x 10**9/L
  * Hemoglobin (Hgb) ≥ 9 g/dL
  * Platelets > 100 x 10**9/L
  * Creatinine ≤ 1.6 mg/dL
  * ALT and AST ≤ 2.5 x ULN
  * Alkaline phosphatase ≤ 5 ULN
  * Total bilirubin ≤ 1.5 mg/dL
* Baseline LVEF ≥ 55% measured by echocardiogram or MUGA scan
* Negative β-HCG pregnancy test (serum) for premenopausal women of reproductive capacity (those who are biologically capable of having children) and for women less than 12 months after the menopause. All subjects who are biologically capable of having children must agree and commit to the use of a reliable method of birth control from 2 weeks before administration of the first dose of investigational product until 28 days after the last dose of investigational product
* Absence of any psychological, familial, sociological, or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial

Exclusion Criteria:

* Clinical or radiologic evidence of metastatic disease at the time of study entry
* Prior chemotherapy, radiotherapy, or surgery for BC, other than excision of a tumor in the contralateral breast, and provided that the patient did not previously receive adjuvant radiotherapy or chemotherapy
* Subjects with a concurrently active second malignancy, other than adequately treated non melanoma skin cancers, in situ melanoma or in situ cervical cancer. Subjects with other non-mammary malignancies must have been disease-free for at least 5 years
* Known or suspected hypersensitivity reaction to any investigational or therapeutic compound or their incorporated substances
* Presence of CHF or LVEF < 55%
* Clinically significant (i.e. active) cardiovascular disease, including cerebrovascular accident (< 6 months before enrollment), unstable angina pectoris, myocardial infarction ≤ 6 months before enrollment, uncontrolled hypertension (systolic > 150 mmHg and/or diastolic > 100 mmHg), or high-risk uncontrolled arrhythmias
* Uncontrolled diabetes mellitus, active peptic ulcer disease, or uncontrolled epilepsy
* Active uncontrolled infection at the time of enrolment
* History of significant co-morbidities that, in the judgment of the investigator, may interfere with the conduction of the study, the evaluation of response, or with informed consent
* Use of any investigational agent or participation in another therapeutic clinical trial concurrently or in the previous 30 days before the enrollment
* Patients who are pregnant or breast-feeding
* Women of child-bearing potential who are unable or unwilling to use acceptable contraceptive measures
* Inability or unwillingness to abide by the study protocol or cooperate fully with the investigator or designee

Ages: 18 Years to 74 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2013-06; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Rate of symptomatic (type A) and asymptomatic (type B) cardiac events during the study treatment period | Following 12 months after first dose of the study treatment

SECONDARY OUTCOMES:
pCR in breast (pCRB) | At the time of definitive surgery, an expected average of 23 weeks
pCR in breast and axilla (pCRBA) | At the time of definitive surgery, an expected average of 23 weeks
Clinical objective response rate (cORR) in the breast and axilla by RECIST criteria version 1.1 | At the time of definitive surgery, an expected average of 23 weeks
Residual Cancer Burden (RCB) at surgery following the procedures of the MD Anderson Cancer Center | At the time of definitive surgery, an expected average of 23 weeks
Breast conservation rate at surgery | At the time of definitive surgery, an expected average of 23 weeks
Evaluation of serum biomarkers predictive of cardiotoxicity | Following 12 months after first dose of the study treatment
Percentage of patients with grade 3/4 neutropenia (assessed by CTCAE v.4) | Following 12 months after first dose of the study treatment
Time of onset and time of recovery from symptomatic (type A) and asymptomatic (type B) cardiac events (assessed by CTCAE v.4) | Following 12 months after first dose of the study treatment
Dose reductions due to treatment toxicity (assessed by CTCAE v.4) | Following 12 months after first dose of the study treatment
Dose delays due to treatment toxicity (assessed by CTCAE v.4) | Following 12 months after first dose of the study treatment
Number of patients with adverse events and serious adverse events (assessed by CTCAE v.4) | Following 12 months after first dose of the study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Joaquín Gavilá Gregori, MD, Principal Investigator — Fundación Instituto Valenciano de Oncología
Locations (19):
- Spain (19):
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Universitario Vall d´Hebron, Barcelona
  - Complejo Hospitalario San Pedro de Alcántara, Cáceres
  - Hospital Universitari Arnau de Vilanova de Lleida, Lleida
  - Hospital Universitario 12 de Octubre, Madrid
  - Centro Integral Oncológico Clara Campal, Madrid
  - Hospital Universitario Clínico San Carlos, Madrid
  - Hospital Universitario Puerta de Hierro de Majadahonda, Madrid
  - MD Anderson Cancer Center Madrid, Madrid
  - Hospital Universitario Virgen de la Arrixaca, Murcia
  - Hospital Son Llàtzer, Palma de Mallorca
  - Hospital Universitari Son Espases, Palma de Mallorca
  - Hospital Sant Joan de Reus, Reus
  - Hospital Sagrado Corazón USP, Seville
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Virgen de la Macarena, Seville
  - Fundación Instituto Valenciano de Oncología, Valencia
  - Hospital Arnau de Vilanova de Valencia, Valencia
  - Hospital Universitario Lozano Blesa, Zaragoza

REFERENCES:
- [Background] Gavilá J, Llombart A, Guerrero A, Ruíz A, Climent M, Guillem V. Opti-HER HEART: A prospective, multicenter, single-arm, phase II study to evaluate the safety of neoadjuvant liposomal doxorubicin plus paclitaxel, trastuzumab, and pertuzumab in patients with operable HER2-positive breast cancer. Poster session presented at: 35th Annual San Antonio Breast Cancer Symposium (SABCS); 2012 December 4th-8th; San Antonio, Texas, United States.
- [Derived] Gavila J, Oliveira M, Pascual T, Perez-Garcia J, Gonzalez X, Canes J, Pare L, Calvo I, Ciruelos E, Munoz M, Virizuela JA, Ruiz I, Andres R, Perello A, Martinez J, Morales S, Marin-Aguilera M, Martinez D, Quero JC, Llombart-Cussac A, Prat A. Safety, activity, and molecular heterogeneity following neoadjuvant non-pegylated liposomal doxorubicin, paclitaxel, trastuzumab, and pertuzumab in HER2-positive breast cancer (Opti-HER HEART): an open-label, single-group, multicenter, phase 2 trial. BMC Med. 2019 Jan 9;17(1):8. doi: 10.1186/s12916-018-1233-1. PMID 30621698
- See also: SOLTI Breast Cancer Research Group — http://www.gruposolti.org